CLINICAL TRIAL: NCT03265860
Title: Intravoxel Incoherent Motion Prognostic Value in the Initial Evaluation of Patients With Acute Ischemic Strokes Using 3 Tesla Magnetic Resonance Imaging
Acronym: IMPROVES
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2017_5
Record Dates: First submitted 2017-08-28; First posted 2017-08-29 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Magnetic Resonance Imaging
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IntraVoxel Incoherent Motion sequence — The IVIM diffusion sequence with a duration of 2 minutes is added to the imaging protocol.

SUMMARY:
Ischemic strokes are the first cause of handicap in adult people, the second cause of dementia and the third cause of death in France. Brain Magnetic Resonance (MR) initial assessment is mandatory to get the right diagnosis, to exclude hemorrhagic lesions and to determine the best treatment.

The conventional diffusion weighted imaging sequence is used to establish the diagnosis and to estimate the volume of ischemic lesions. The perfusion weighted imaging sequences are also used to assess the diffusion-perfusion mismatch which is supposed to be the ischemic penumbra corresponding to territories that could be saved with appropriate treatments.

IntraVoxel Incoherent Motion (IVIM) is a multi-b diffusion sequence which allows to extract four quantitative variables (D, D*, f, ADC) related to the true molecular diffusion and correlated to the microvascular perfusion.

It's a quick sequence with no need of contrast injection and allowing a perfect coregistration with the true diffusion. It has been validated in many pathologies but not in acute strokes.

The feasibility of this sequence in acute ischemic strokes has already been assessed with interesting results.

The study aims to assess the correlation between the quantitative values of IVIM at initial MR exam and the modified Rankin Scale (mRS) score 3 months after an acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Admitted for an acute ischemic stroke
* Affiliated to a Social Security scheme

Exclusion Criteria:

* Absolute contraindications to MRI
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Correlation between quantitative values of IntraVoxel Incoherent Motion at initial Magnetic Resonance Imaging (MRI) and the modified Rankin Scale (mRS) at 3 months after an acute ischemic stroke. | 3 months
  IntraVoxel Incoherent Motion is a diffusion sequence which allows to extract four quantitative variables (D, D*, f, ADC) related to the true molecular diffusion and correlated to the microvascular perfusion.
  We aim to assess the correlation between the quantitative values of IVIM at initial exam and the mRS score 3 months after an acute ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Augustin Lecler, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided